CLINICAL TRIAL: NCT05800743
Title: Evaluation of the GORE® Ascending Stent Graft in the Treatment of Lesions of the Ascending Aorta
Brief Title: Evaluation of the GORE® Ascending Stent Graft
Acronym: ARISEII
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASG 22-02
Record Dates: First submitted 2023-03-23; First posted 2023-04-06 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Aortic Aneurysm, Thoracic; Pseudoaneurysm; Aortic Dissection; Aorta; Lesion
Keywords: Ascending Aorta; Pseudoaneurysm; Aortic Lesion; Endovascular Repair; Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aneurysm, False; Aortic Dissection | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- ASG device only in Ascending Aorta (Experimental): Ascending Aortic Isolated Lesions, Pseudoaneurysms and Penetrating Aortic Ulcers in subjects at high-risk for surgical repair, treated with endovascular repair using the ASG device alone.
  Interventions: Device: GORE® Ascending Stent Graft (ASG device)
- ASG + TBE (Experimental): Ascending Aorta/Aortic Arch Isolated Lesions and Chronic De Novo Dissections in subjects at high-risk for surgical repair, treated with endovascular repair using the ASG and TBE devices.
  Interventions: Device: GORE® Thoracic Aortic Graft Thoracic Branch Endoprosthesis (TBE Device)
- Surgical Follow-up Cohort (Other): Open surgical repair of ascending aorta in subjects at high-risk for surgical repair
  Interventions: Procedure: Surgery

INTERVENTIONS:
Device: GORE® Ascending Stent Graft (ASG device) — Endovascular aortic repair of the ascending aorta
  Arms: ASG device only in Ascending Aorta
Device: GORE® Thoracic Aortic Graft Thoracic Branch Endoprosthesis (TBE Device) — Endovascular aortic repair of the ascending aorta/aortic arch
  Other Names: Revascularization Procedure
  Arms: ASG + TBE
Procedure: Surgery — Open surgical repair of the ascending aorta and/or the aortic arch
  Arms: Surgical Follow-up Cohort

SUMMARY:
The primary objective of ARISE II is to assess the safety and effectiveness of the GORE® Ascending Stent Graft device in the treatment of lesions involving the ascending aorta and aortic arch.

ELIGIBILITY:
Inclusion Criteria: ASG Device Alone Arm

The patient is/has:

1. Ascending Aortic pathologies warranting surgical repair compatible with the treatment requirements of the ASG device meeting any of the following criteria: Aneurysm

   1. Fusiform aneurysm (≥50mm or documented growth rate >0.5cm/year)
   2. Saccular aneurysm (no diameter criteria)
   3. Pseudoaneurysms (>30 days post-surgery, no diameter criteria) Non-aneurysm
   4. Penetrating Aortic Ulcers (PAUs) (no diameter criteria)
   5. Pseudoaneurysms, following open surgical repair of a Type A dissection (>30 days post-surgery, no diameter criteria)
2. Anatomic compatibility with ASG device based on Gore Imaging Sciences review.

   1. Treatment must be limited to the ascending aorta
   2. Lesion location is ≥2cm distal to the most distal coronary artery ostia
   3. Distal extent of the lesion is located ≥2cm proximal to the origin of the Brachiocephalic Artery (BCA)
   4. Proximal and distal landing zones must be ≥2cm in length
   5. Landing zones cannot be heavily calcified, or heavily thrombosed
   6. Landing zone diameter between 27mm - 48mm
   7. For patients with prior replacement of the ascending aorta and/or aortic arch by an endovascular or surgical graft, there must be at least ≥2 cm overlap of ASG device and previously implanted graft.
3. Considered high-risk for open surgical repair by meeting any of the following criteria:

   1. ≥75 years of age
   2. Previous median sternotomy
   3. Documented identification of other subject-specific risk factors (e.g., medical history, active medical diagnosis) by a study investigator and an experienced open ascending and/or aortic arch surgeon (e.g., cardiothoracic surgeon).
4. Age ≥18 years at time of informed consent signature
5. Adequate vascular access via transfemoral or retroperitoneal approach
6. Informed Consent Form (ICF) signed by the subject or legally authorized representative
7. Agrees to comply with protocol requirements, including imaging and 5-year follow-up

Exclusion Criteria: ASG Device Alone Arm

The patient is/has:

1. De novo Type A dissection
2. Requires immediate treatment
3. Dissected great vessels requiring treatment
4. Anticipated need for coronary or aortic valve intervention within one year post treatment
5. Any aortic valve repair or replacement including transcatheter aortic valve replacement (TAVR) or coronary artery intervention within 30 days prior to treatment
6. Complex percutaneous coronary intervention (PCI) or treatment for acute coronary syndrome requiring Dual Anti Platelet Therapy (DAPT) within 30 days prior to treatment
7. Open chest surgical repair within 30 days prior to treatment
8. Presence of Intramural Hematoma (IMH) in landing zones
9. Prosthetic heart valve in the aortic position that precludes safe delivery of the ASG device
10. Aortic insufficiency grade 3 or greater
11. Previous endovascular repair with a non-Gore device that would interfere with or result in contact with planned repair
12. Concomitant vascular disease requiring treatment that is not planned for index endovascular procedure
13. Any stroke or myocardial infarction within 6 weeks prior to treatment
14. Presence of protruding and/or irregular thrombus and/or atheroma in the ascending aorta or aortic arch or any other factors that could increase the risk of stroke based on imaging review
15. Known degenerative connective tissue disease (e.g., Marfan's or Ehler-Danlos Syndrome, EDS)
16. Participation in investigational drug or medical device study within one year of enrollment unless approved by the sponsor
17. Known history of drug abuse within one year of treatment
18. Pregnant at time of procedure
19. Active infected aorta, mycotic aneurysm
20. Active systemic infection (e.g., infection requiring treatment with parenteral anti-infective medication)
21. Renal failure, defined as patients with an estimated Glomerular Filtration Rate (eGFR) <30 (mL/min/1.73 m2) or currently requiring dialysis
22. Life expectancy <12 months
23. Known sensitivities or allergies to the device materials
24. Known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment
25. Body habitus or other medical condition which prevents adequate fluoroscopic and CT visualization of the aorta

Inclusion Criteria: ASG + TBE Device Arm

The patient is/has:

1. Ascending and/or Arch Aortic pathologies warranting surgical repair compatible with the treatment requirements of the ASG device and meeting any of the following criteria: Aneurysms

   1. Fusiform aneurysm (≥55 mm or documented growth rate >0.5cm/year)
   2. Saccular aneurysm (no diameter criteria)
   3. Pseudoaneurysms (>30 days post-surgery, no diameter criteria) Non-aneurysms
   4. Penetrating Aortic Ulcers (no diameter criteria)
   5. Pseudoaneurysms, following open surgical repair of a Type A dissection (>30 days post-surgery, no diameter criteria)
   6. Chronic de novo (>90 days) Type A aortic dissection requiring treatment

      * Chronic de novo aortic dissection with primary entry tear in the ascending aorta or arch
      * Chronic de novo aortic dissection with primary entry tear in the descending thoracic aorta with retrograde involvement of the aortic arch and/or ascending aorta
   7. Residual aortic dissection following surgical repair of Type A aortic dissection requiring treatment (>30 days post-surgery)
2. Anatomic compatibility with ASG device used in combination with the TBE Device based on Gore Imaging Sciences review.

   Proximal Aortic Landing Zone:
   1. Landing zone is native aorta or surgical graft
   2. Lesion location is ≥2cm distal to the most distal coronary artery ostia
   3. Proximal landing zone must be ≥2cm in the ascending aorta.
   4. Landing zone cannot be aneurysmal, heavily calcified, or heavily thrombosed
   5. Landing zone diameter between 27mm - 48mm
   6. Acceptable proximal landing zone outer curvature length for the required device

   Branch Vessel Landing Zone:
   1. Length of ≥2.5 cm proximal to first major branch vessel
   2. Target branch vessel inner diameters of 11-18 mm
   3. Target branch vessel landing zone must be in native vessel that cannot be heavily calcified, or heavily thrombosed

   Distal Aortic Landing Zone:
   1. Outer curvature must be ≥2 cm proximal to the celiac artery
   2. Aortic inner diameters between 16-42 mm
   3. Landing zone in native aorta or previously implanted GORE® TAG® Conformable Thoracic Stent Graft (CTAG Device)
3. Considered high-risk for open surgical repair by meeting any of the following criteria:

   1. ≥75 years of age
   2. Previous median sternotomy
   3. Documented identification of other subject-specific risk factors (e.g., medical history, active medical diagnosis) by a study investigator and an experienced open ascending and/or aortic arch surgeon (e.g., cardiothoracic surgeon).
4. Age ≥18 years at time of informed consent signature
5. Adequate vascular access via transfemoral or retroperitoneal approach
6. Informed Consent Form (ICF) signed by the subject or legally authorized representative
7. Agrees to comply with protocol requirements, including imaging and 5-year follow-up

Exclusion Criteria: ASG + TBE Device Arm

The patient is/has:

1. Acute and subacute de novo Type A dissection (defined as <90 days)
2. Requires immediate treatment
3. Dissected great vessels requiring treatment
4. Anticipated need for coronary or aortic valve intervention within one year post treatment
5. Any aortic valve repair or replacement including transcatheter aortic valve replacement (TAVR) or coronary artery intervention within 30 days prior to treatment
6. Complex percutaneous coronary intervention (PCI) or treatment for acute coronary syndrome requiring Dual Anti Platelet Therapy (DAPT) within 30 days prior to treatment.
7. Open chest surgical repair within 30 days prior to treatment
8. Presence of Intramural Hematoma (IMH) in landing zones
9. Prosthetic heart valve in the aortic position that precludes safe delivery of the ASG device
10. Aortic insufficiency grade 3 or greater.
11. Previous endovascular repair with a non-Gore device that would interfere with or result in contact with planned repair
12. Concomitant vascular disease requiring treatment that is not planned for index endovascular procedure
13. Any stroke or myocardial infarction within 6 weeks prior to treatment
14. Presence of protruding and/or irregular thrombus and/or atheroma in the ascending aorta or aortic arch or any other factors that could increase the risk of stroke based on imaging review
15. Known degenerative connective tissue disease (e.g., Marfan Syndrome or Ehlers-Danlos Syndrome, EDS)
16. Participation in investigational drug or medical device study within one year of enrollment unless approved by the sponsor
17. Known history of drug abuse within one year of treatment
18. Pregnant at time of procedure
19. Active infected aorta, mycotic aneurysm
20. Active systemic infection (e.g., infection requiring treatment with parenteral anti-infective medication)
21. Renal failure, defined as patients with an estimated Glomerular Filtration Rate (eGFR) <30 (mL/min/1.73 m2) or currently requiring dialysis
22. Life expectancy <12 months
23. Known sensitivities or allergies to the device materials
24. Known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment
25. Body habitus or other medical condition which prevents adequate fluoroscopic and CT visualization of the aorta
26. Previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or known hypersensitivity to heparin or a history of a hypercoagulability disorder and/or state

Inclusion Criteria: Surgical Follow-up Cohort

Subjects who meet the following criteria will be followed:

1. The aortic lesion involves the ascending aorta and/or aortic arch
2. The subject is determined to be high-risk for open surgical repair per the protocol requirements
3. The subject is at least 18 years of age
4. The subject is willing to comply with the protocol requirements
5. Open surgery to repair the aortic lesion the patient was screened for is intended to be performed at the investigational site responsible for initiating the screening process for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Primary effectiveness endpoint as measured by device technical success and absence of reintervention. | 30 Days
  The primary effectiveness endpoint is a composite of the following events through one month post procedure: Device Technical Success and Absence of Reintervention.
  Technical Success is defined as including:
  1. Successful access and delivery to the intended implantation site, and retrieval of the device delivery system, and;
  2. Accurate placement of the device at the intended implantation site, and
  3. Patency of the graft in absence of clinically significant device deformations (e.g., kinking, stent eversion, mal-deployment, misaligned deployment), and
  Absence of reintervention is defined as: The absence of unanticipated additional procedures related to the device, procedure, or withdrawal of the delivery system
Primary Safety Endpoint as measured by a composite of the absence of aortic rupture, lesion-related mortality, disabling stroke, permanent paraplegia, permanent paraparesis, and new onset renal failure requiring permanent dialysis. | 30 Days
  The primary safety endpoint is a composite of the following events through 30 days post endovascular procedure:
  * Aortic rupture
  * Lesion-related mortality
  * Disabling Stroke
  * Permanent paraplegia
  * Permanent paraparesis
  * New onset renal failure requiring permanent dialysis

SECONDARY OUTCOMES:
Secondary endpoints as measured as a composite of procedural and treatment success. | 30 Days, and 6, 12, 24, 36, 48 and 60 months
  Two secondary endpoints are planned for the study with no inferential analysis. Composite endpoint of procedural success elements measured at one month follow-up Composite endpoint of treatment success elements measured at all appropriate follow-up windows
Secondary endpoint as measured by Short Form-36® physical component summary (PCS) | 12 months
  Short Form-36® PCS measured at the one year follow-up visit with inferential analysis

CONTACTS AND LOCATIONS:
Overall Officials: Eric Roselli, MD, Principal Investigator — The Cleveland Clinic
Locations (39):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - MemorialCare Heart and Vascular Institute - Long Beach Medical Center, Long Beach, California
  - Keck Medical Center University of Southern California, HCC II, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford Hospital, Stanford, California
  - University of Colorado Hospital Authority, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida - Gainesville, Gainesville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University -Bluhm Cardiovascular Institute, Clinical Trials Unit, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Frankel Cardiovascular Center, Ann Arbor, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine - St. Louis, St Louis, Missouri
  - Hackensack UMC, Hackensack, New Jersey
  - Westchester Medical Center, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OhioHealth Research and Innovation Institute, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Methodist DeBakey Heart & Vascular Center, Houston, Texas
  - The Heart Hospital at Baylor Plano, Plano, Texas
  - Intermountain Heart Institute, Murray, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Sentara Mid Atlantic Cardiothoracic Surgeons, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - West Virginia University Medicine, Morgantown, West Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin